CLINICAL TRIAL: NCT04551742
Title: Social & Contextual Impact on Children Undergoing Liver Transplantation
Acronym: SOCIAL-TX
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 19-29632
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplantation; Liver Diseases
Keywords: Pediatric; Health services research; Social determinants of health
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The social determinants of health have a large impact on health. For example, neighborhood socioeconomic deprivation is associated with increased risk of medication non-adherence, graft failure, and death in children after liver transplant. In order to address these socioeconomic inequities in outcomes, a more granular understanding of how the social determinants of health impact outcomes is needed. In this observational prospective cohort, caregivers of children undergoing liver transplantation will complete surveys and undergo in-depth, qualitative interviews. The survey will assess comprehensively for the social determinants of health (e.g. material economic hardship, health literacy, social connectedness, primary care quality, etc). The qualitative interviews will identify barriers and facilitators that socioeconomically deprived children/families have to obtaining the ideal outcome and identify health system opportunities to integrate social needs and medical care. Data will be linked to an existing prospective cohort study (The Society for Pediatric Liver Transplant registry) to assess the impact of social risk on outcomes after transplant.

Healthcare providers who take care of children undergoing liver transplant will also be included in the qualitative interviews. The goal of including this group in the study is to determine the health systems barriers and facilitators to social needs screening and intervention.

ELIGIBILITY:
Inclusion Criteria:

Caregivers/parents of children with the following criteria will be approached for inclusion in this study:

* Children <18 years of age at the time of transplant
* Undergoing liver transplantation
* Guardian's consent, child assent (in accordance with each institution's IRB policies)
* Consents to enrollment in SPLIT

Exclusion Criteria:

Caregivers/parents of children undergoing liver transplantation will be excluded it:

* Caregiver unwilling or unable to complete the survey
* Child is a ward of the state (e.g., foster care) since present circumstances may not be reflective of child's past or future circumstances
* Non-English, non-Spanish speakers
* Non-US residents
* Declined participation in SPLIT

Inclusion Criteria for Interview Portion of the Study:

* Participants who have completed the questionnaire OR
* Medical team member involved in the care of children undergoing liver transplant (e.g., physician, nurse, social worker)

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Caregivers or parents of children undergoing liver transplantation Healthcare professionals caring for children undergoing liver transplantation
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of days hospitalized within 90 days after transplant, including the initial transplant hospitalization | 90 Days
Episodes of acute cellular rejection | 1 Year
Ideal Outcome-3 (IO-3) | 3 Years
  The ideal outcome measure is a composite measure of morbidity after transplant defined as alive, ALT and GGT <50, normal GFR, no non-liver transplants, no cytopenias, and no PTLD.

SECONDARY OUTCOMES:
Readmission within 90 days after transplant | 90 Days
Episode of biopsy-proven acute cellular rejection within 90 days after transplant | 90 Days
Episode of re-transplantation | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Sharad Wadhwani, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (8):
- United States (8):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No